CLINICAL TRIAL: NCT07407036
Title: Electromyographic and Functional Analysis of Neuromuscular Rehabilitation Methods in Individuals With Scapholunate Instability: A Comparison of Conventional and Virtual Reality-Supported Interventions
Brief Title: Conventional and Virtual Reality-Based Neuromuscular Rehabilitation in Scapholunate Instability
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Yeditepe University (Other)
Collaborators: Biruni University (Other); Scientific and Technological Research Council of Turkey (TÜBİTAK) (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Eda1
Record Dates: First submitted 2026-02-05; First posted 2026-02-12 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Scapholunate Instability
Keywords: Scapholunate Instability; Wrist Proprioception; Surface Electromyography; Neuromuscular Rehabilitation

STUDY DESIGN:
Intervention Model Description: Participants will be randomly assigned to one of two parallel groups: a conventional physiotherapy group or a virtual reality-supported neuromuscular rehabilitation group. Randomization will ensure that participants have an equal chance of being allocated to either group. Each participant will be assigned to a single study arm for the entire duration of the study and will not cross over to the other group. Both groups will receive conventional physiotherapy, while the intervention group will additionally receive virtual reality-supported neuromuscular rehabilitation. Both interventions will be delivered over an 8-week period with the same treatment frequency. Outcomes will be assessed before and after the intervention, and between-group comparisons will be performed to evaluate the effects of the two rehabilitation approaches.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional Physiotherapy Group (Active Comparator): Participants assigned to this arm will receive a structured conventional physiotherapy program focusing on wrist and forearm stabilization. The intervention will include strengthening exercises targeting scapholunate-friendly muscles, neuromuscular control exercises, and proprioceptive training aimed at improving wrist stability and functional movement patterns. The program will be delivered under supervision twice per week for 8 weeks.
  Interventions: Other: Conventional Physiotherapy Group
- Virtual Reality-Supported Neuromuscular Rehabilitation Group (Experimental): Participants assigned to this arm will receive the same conventional physiotherapy program as the control group. In addition, they will participate in virtual reality-supported neuromuscular rehabilitation using sensor-based interactive therapeutic games designed for upper extremity rehabilitation. The virtual reality component will consist of four different game-based tasks targeting wrist and forearm motor control, proprioceptive feedback, and functional task performance. These games will be selected to promote controlled movement, coordination, and task-oriented motor training. The intervention will be administered twice per week for 8 weeks under physiotherapist supervision.
  Interventions: Other: Conventional Physiotherapy Group; Other: Virtual Reality-Supported Neuromuscular Rehabilitation

INTERVENTIONS:
Other: Conventional Physiotherapy Group — Participants assigned to the conventional physiotherapy group will receive a structured neuromuscular rehabilitation program focusing on wrist and forearm stabilization. The intervention will include supervised strengthening exercises targeting scapholunate-friendly muscles, neuromuscular control exercises, and proprioceptive training aimed at improving wrist stability and functional movement patterns. Progressive resistance and task-oriented exercises will be used according to individual tolerance. The rehabilitation program will be administered twice per week for 8 weeks by a licensed physiotherapist.
Other: Virtual Reality-Supported Neuromuscular Rehabilitation — Participants in the virtual reality-supported rehabilitation group will receive the same conventional physiotherapy program as the control group. In addition, this group will participate in virtual reality-based therapeutic exercises delivered through sensor-based interactive games designed for upper extremity rehabilitation. These exercises will aim to enhance wrist and forearm motor control, proprioceptive feedback, and functional task performance by promoting controlled and task-oriented movement patterns. Virtual reality sessions will be supervised by a physiotherapist and integrated into the rehabilitation program with the same frequency and duration as the conventional intervention, administered twice per week over an 8-week period.
  Arms: Virtual Reality-Supported Neuromuscular Rehabilitation Group

SUMMARY:
Scapholunate instability is a common form of carpal instability that can cause wrist pain, weakness, and functional limitations during daily activities. Conservative rehabilitation approaches are frequently recommended in the early stages; however, there is no standardized rehabilitation protocol, and the effects of different neuromuscular rehabilitation methods have not been sufficiently investigated.

The primary aim of this study is to comparatively examine the effects of conventional physiotherapy approaches and virtual reality-supported neuromuscular rehabilitation on forearm muscle activation patterns assessed using surface electromyography, wrist proprioceptive function (joint position sense), pain intensity, and functional improvement in individuals with scapholunate instability, and to identify clinically applicable rehabilitation protocol approaches for this population.

In this single-blind randomized controlled trial, participants with pre-dynamic or dynamic scapholunate instability will be randomly assigned to either a conventional rehabilitation group or a virtual reality-supported rehabilitation group. Both groups will receive an 8-week rehabilitation program administered twice per week. Primary outcome measures will include electromyographically assessed forearm muscle activation and wrist proprioception. Secondary outcome measures will include pain intensity, grip strength, wrist muscle strength, and upper extremity functional outcomes assessed using validated clinical instruments. All outcome assessments will be performed before and after the intervention period by an assessor blinded to group allocation.

DETAILED DESCRIPTION:
Scapholunate instability is the most common form of carpal instability and is characterized by disruption of the scapholunate interosseous ligament, leading to altered wrist kinematics, pain, reduced grip strength, proprioceptive deficits, and functional limitations. In the early (pre-dynamic and dynamic) stages of the condition, conservative management is recommended; however, standardized, evidence-based rehabilitation protocols are lacking. In particular, the neuromuscular mechanisms underlying wrist stabilization, muscle activation patterns, and proprioceptive control have not been sufficiently investigated using objective measurement methods.

This randomized, single-blinded controlled trial is designed to compare the effects of conventional physiotherapy and virtual reality-supported neuromuscular rehabilitation in individuals with scapholunate instability. Participants diagnosed with pre-dynamic or dynamic scapholunate instability will be randomly allocated to either a conventional rehabilitation group or a virtual reality-supported rehabilitation group. Both groups will receive an 8-week intervention program consisting of two supervised sessions per week. The conventional rehabilitation program will focus on strengthening "scapholunate-friendly" wrist and forearm muscles, improving neuromuscular control, and enhancing wrist proprioception through progressive strengthening and proprioceptive exercises. The intervention group will receive the same conventional program supplemented with virtual reality-based rehabilitation games designed to promote task-oriented movement, sensorimotor integration, and real-time feedback.

Outcome assessments will be conducted before and after the intervention by a blinded evaluator. Primary outcome measures will include wrist proprioception (joint position sense) and forearm muscle activation patterns assessed using surface electromyography. Secondary outcome measures will include pain intensity, grip strength, wrist muscle strength, pressure pain threshold, and upper extremity functional performance assessed using validated clinical outcome measures.

The study aims to objectively evaluate neuromuscular and proprioceptive changes associated with different rehabilitation approaches and to determine whether virtual reality-supported rehabilitation provides additional benefits over conventional physiotherapy alone. The findings of this study are expected to contribute to the development of clinically applicable, evidence-based rehabilitation protocols for individuals with scapholunate instability and to provide insight into muscle activation strategies involved in wrist stabilization.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 18 and 65 years
* Diagnosed with scapholunate instability (pre-dynamic or dynamic instability) by a physician and referred for conservative treatment
* A score of ≤6 on the Beighton Hypermobility Scale
* Presence of clinical instability symptoms, including pain, a sense of instability, and functional limitation
* Willingness to participate in the study and high motivation to comply with the intervention protocol

Exclusion Criteria:

* History of previous surgery involving the hand or wrist
* Presence of any neurological or cardiovascular disorder
* Presence of additional orthopedic pathology affecting the shoulder, elbow, or wrist other than scapholunate instability
* History of surgery involving the ipsilateral upper extremity within the past 6 months
* Presence of visual or hearing impairments that may interfere with participation in the rehabilitation program
* Participation in sensory- or function-oriented rehabilitation of either hand within the past 6 months
* A score below 26 on the Montreal Cognitive Assessment (MoCA)
* Inability to read or write

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-03 (Estimated); Primary Completion 2026-12 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Wrist Proprioception | Baseline and after 8 weeks of intervention
  Wrist proprioception will be assessed by evaluating joint position sense using both a universal goniometer and an electrogoniometer. Assessments will be performed in a standardized sitting position with the forearm supported. Predetermined wrist joint angles will be set by the assessor, and participants will be asked to actively reproduce the target positions without visual feedback. Wrist joint angles will be recorded using both measurement tools, and the absolute angular error between the target angle and the reproduced angle will be calculated to determine proprioceptive accuracy.
Forearm Muscle Activation | Baseline and after 8 weeks of intervention
  Forearm muscle activation will be assessed using surface electromyography during standardized wrist and forearm tasks. Electromyographic activity of selected forearm muscles involved in wrist stabilization will be recorded and analyzed to evaluate neuromuscular activation patterns.

SECONDARY OUTCOMES:
Pain Intensity | Baseline and after 8 weeks of intervention
  Pain intensity will be assessed using the Visual Analog Scale (VAS). Participants will rate their wrist pain on a 10-cm horizontal line, where higher scores indicate greater pain intensity.
Pressure Pain Threshold | Baseline and after 8 weeks of intervention
  Pressure pain threshold will be measured using a pressure algometer applied to predefined and standardized anatomical sites around the wrist. Gradually increasing pressure will be applied perpendicular to the skin at a constant rate, and participants will be instructed to indicate the point at which the sensation first becomes painful. The pressure value at this point will be recorded as the pressure pain threshold, with higher values indicating lower pain sensitivity.
Grip Strength | Baseline and after 8 weeks of intervention
  Grip strength will be measured using a hand dynamometer under standardized testing conditions. Participants will be seated with the shoulder adducted, elbow flexed at 90 degrees, and the forearm in a neutral position. Each participant will be instructed to perform a maximum voluntary grip contraction. Three consecutive measurements will be taken, and the highest value will be recorded to evaluate changes in hand strength.
Wrist Muscle Strength | Baseline and after 8 weeks of intervention
  Wrist muscle strength will be assessed using standardized strength testing of wrist flexion, extension, radial deviation, and ulnar deviation. Strength measurements will be performed in a standardized sitting position with the forearm supported, and resistance will be applied manually by the assessor. Participants will be instructed to perform maximum voluntary contractions for each movement, and the obtained strength values will be recorded to evaluate changes in wrist strength following the intervention.
Upper Extremity Function (QuickDASH) | Baseline and after 8 weeks of intervention
  Upper extremity function and symptoms will be evaluated using the Quick Disabilities of the Arm, Shoulder and Hand (QuickDASH) questionnaire. This self-reported outcome measure consists of 11 items assessing physical function and symptoms related to upper extremity activities. Participants will rate their level of difficulty in performing daily activities over the previous week. Scores range from 0 to 100, with higher scores indicating greater disability.
Wrist Pain and Disability (PRWE) | Baseline and after 8 weeks of intervention
  Wrist-specific pain and disability will be assessed using the Patient-Rated Wrist Evaluation (PRWE) questionnaire. The PRWE is a self-reported instrument consisting of pain and function subscales that evaluate wrist-related pain intensity and functional difficulty during daily activities. Participants will complete the questionnaire based on their symptoms over the previous week. Scores range from 0 to 100, with higher scores indicating greater wrist pain and functional disability.

CONTACTS AND LOCATIONS:
Overall Officials: Zeynep HOSBAY, Professor, Principal Investigator — Biruni University, Faculty of Health Sciences, Department of Physiotherapy and Rehabilitation
Locations (1):
- Biruni University, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No